CLINICAL TRIAL: NCT02770248
Title: 24-hr Intraocular Pressure Control With Brinzolamide 1% / Brimonidine 0.2% Ophthalmic Suspension vs Vehicle
Brief Title: 24-hr Intraocular Pressure Control With SIMBRINZA ®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLT320a-P001
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Results first posted 2018-01-04 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-01

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — brinzolamide; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIMBRINZA (Experimental): Brinzolamide 1% / Brimonidine 0.2% tartrate ophthalmic suspension, 1 drop 3 times per day in each eye at 8 AM, 3 PM, and 10 PM for 28 days
  Interventions: Drug: Brinzolamide 1%/brimonidine 0.2% tartrate ophthalmic suspension
- Vehicle (Active Comparator): Vehicle, 1 drop 3 times per day in each eye at 8 AM, 3 PM, and 10 PM for 28 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine 0.2% tartrate ophthalmic suspension
  Other Names: SIMBRINZA ®
  Arms: SIMBRINZA
Drug: Vehicle — Inactive ingredients used as a placebo for masking purposes
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate differences between treatments in mean change from baseline in 24-hr intraocular pressure (IOP) at Week 4.

DETAILED DESCRIPTION:
Subjects will undergo washout of pre-study IOP-lowering medications for the appropriate duration, then undergo 2 eligibility visits. Eligible subjects will be randomized 1:1, to receive masked SIMBRINZA ® or Vehicle for 4 weeks. Two 24-hour visits will be conducted (Day 0 and Week 4) during which intraocular pressure will be collected every 2 hours. The expected duration of subject participation in the study is 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either open-angle glaucoma or ocular hypertension;
* Able to attend all study related visits and be housed overnight at clinical site for the study assessments;
* Willing and able to sign an informed consent form;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential who are pregnant, intend to become pregnant during the study, breast-feeding, or not using adequate birth control;
* Diagnosed with any form of glaucoma other than open angle glaucoma or ocular hypertension;
* Ocular surgeries or procedures excluded by the protocol;
* Diseases, illnesses, infections, or ocular abnormalities excluded by the protocol;
* Best-corrected visual acuity score less than 55 ETDRS letters (equivalent to approximately 20/80 Snellen) in either eye;
* Other protocol-specific exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-01-14 (Actual); Study Completion 2017-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GCRA, Study Director — Alcon Research

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 16 study centers located in the United States.
Pre-assignment Details: Of the 162 enrolled, 37 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (125).
Period: Overall Study
Arm/Group | SIMBRINZA | Vehicle
Started | 62 | 63
Completed | 62 | 61
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Randomized in error, prior to treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who received Investigational Product (IP) and completed at least 1 scheduled on-therapy study visit (Full Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | SIMBRINZA | Vehicle | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (8.52) | 63.6 (11.22) | 65.5 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 41 | 79
  Male | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in 24-hr Intraocular Pressure (IOP) at Week 4
Description: IOP (fluid pressure inside the eye) was measured in millimeters of mercury (mmHg). Change was calculated by taking the change from baseline at each time point and averaging the available changes. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates greater improvement. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 62 | 61
mmHg | -3.09 [-3.6 to -2.5] | -0.60 [-1.2 to -0.1]

2. Secondary Outcome: Least Squares Mean Change From Baseline in Daytime IOP at Week 4
Description: IOP (fluid pressure inside the eye) was measured in mmHg. Change was calculated by taking the change from baseline at each time point (8 AM through 8 PM) and averaging the available changes. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates greater improvement. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 62 | 61
mmHg | -3.93 [-4.5 to -3.3] | -0.51 [-1.1 to 0.1]

3. Secondary Outcome: Least Squares Mean Change From Baseline in Nocturnal IOP at Week 4
Description: IOP (fluid pressure inside the eye) was measured in mmHg. Change was calculated by taking the change from baseline at each time point (10 PM through 6 AM) and averaging the available changes. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates greater improvement. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 62 | 61
mmHg | -1.88 [-2.7 to -1.1] | -0.73 [-1.6 to 0.1]

4. Secondary Outcome: Least Squares Mean Change From Baseline in IOP for Each Time Point (8 AM Through 6 AM) at Week 4
Description: IOP (fluid pressure inside the eye) was measured in mmHg. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates greater improvement. Only one eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Week 4
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | SIMBRINZA | Vehicle
Number analyzed (Participants) | 62 | 61
mmHg
  8AM | -3.28 [-4.0 to -2.5] | -0.49 [-1.2 to 0.3]
  10AM | -5.05 [-5.9 to -4.2] | -0.61 [-1.4 to 0.2]
  12PM | -4.03 [-4.8 to -3.3] | -0.27 [-1.0 to 0.5]
  2PM | -3.36 [-4.2 to -2.5] | -0.66 [-1.5 to 0.2]
  4PM | -3.95 [-4.9 to -3.0] | -0.51 [-1.4 to 0.4]
  6PM | -4.46 [-5.3 to -3.6] | -0.32 [-1.2 to 0.5]
  8PM | -3.42 [-4.3 to -2.5] | -0.72 [-1.6 to 0.2]
  10PM | -2.10 [-3.2 to -1.0] | -0.67 [-1.7 to 0.4]
  12AM | -1.79 [-2.6 to -1.0] | -0.83 [-1.7 to 0.0]
  2AM | -2.30 [-3.4 to -1.2] | -0.55 [-1.7 to 0.6]
  4AM | -1.42 [-2.6 to -0.2] | -0.98 [-2.2 to 0.2]
  6AM | -1.95 [-3.1 to -0.8] | -0.63 [-1.8 to 0.5]

ADVERSE EVENTS:
Time Frame: Day 0 treatment through study completion, an average of 4 weeks
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. Two subjects were administered both Investigational Products. For the Safety analysis, they are grouped under the first administered treatment. "As treated" analysis is reported.
Groups:
- SIMBRINZA: All subjects exposed to SIMBRINZA
- Vehicle: All subjects exposed to Vehicle
Arm/Group | SIMBRINZA | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/64 | 2/60
Other Adverse Events (participants affected / at risk) | 0/64 | 4/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SIMBRINZA (N=64) | Vehicle (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SIMBRINZA (N=64) | Vehicle (N=60)
Conjunctival hyperaemia (Eye disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.